CLINICAL TRIAL: NCT06676748
Title: The Effect of Benzydamine Hydrochloride Spray on Post-operative Sore Throat: a Randomized Controlled Study
Brief Title: Benzydamine Hydrochloride and Post-operative Sore Throat
Acronym: DIFFLAM
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021/2264
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Sore Throat; Postoperative Care
Keywords: Sore throat; Posoperative care; benzydamine hydrochloride; laryngeal mask airway
MeSH Terms: conditions — Pharyngitis | interventions — Benzydamine

STUDY DESIGN:
Intervention Model Description: The study uses a randomized (1:1 allocation ratio) and single-blinded trial design. Block randomization will be used to randomly assign patients to no intervention i.e., usual practice (Control) and BH (Difflam) spray (study) groups in a 1:1 allocation ratio based on a computer-generated code that will be prepared at a remote site and sealed in opaque, sequentially numbered envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Study group will receive Difflam spray by delivering 4 sprays to the posterior pharynx. Patients will be asked to swallow after each spray. Questionnaires will then be administered to the patients 10 minutes after administration of the intervention, and then 4 hours after for their pain scores and side effects, if any.
  Interventions: Drug: Benzydamine Hydrochloride
- Control group (No Intervention): Patients will be asked to fill in questionnaires for their pain scores and side effects, if any.

INTERVENTIONS:
Drug: Benzydamine Hydrochloride — The Difflam Forte Anti-Inflammatory Throat Spray (iNova Pharmaceuticals Pte Ltd, Singapore) is an over-the-counter medication indicated for temporary relief of painful mouth and throat conditions. It contains benzydamine hydrochloride (BH) 3 mg/mL, a non-steroidal anti-inflammatory agent (NSAID), and is recommended for adults to spray 2 to 4 times to the affected throat every 1.5 to 3 hours as needed.
  Other Names: benzydamine hydrochloride 3 mg/mL; Difflam Forte Anti-Inflammatory Throat Spray
  Arms: Study group

SUMMARY:
Postoperative sore throat (POST) after laryngeal mask airway (LMA) insertion is prevalent and unappealing. A significant cause of POST is mechanical injury to the airway mucosa during airway instrumentation, leading to mucosal injury and inflammation. The Difflam Forte Anti-Inflammatory Throat Spray (Difflam) contains benzydamine hydrochloride, a non-steroidal anti-inflammatory agent with topical analgesic properties. This study will randomize 106 women undergoing gynaecological surgery under general anaesthesia with LMA use at KK Women's and Children's Hospital (KKH) in 1:1 allocation ratio of study (Difflam spray) and control (usual practice; no intervention) groups. Demographic and intraoperative airway data collection will be conducted in perioperative period. Those allocated to study group will receive Difflam spray when awake in the post-anaesthesia care unit (PACU). The primary aim to determine if patients undergoing general anaesthesia with LMA use with the Difflam spray in PACU will have a lower incidence of POST in the immediate and 4 hours postoperative recovery period, as compared with those in the control group. Other outcome measures include the severity of pain of sore throat as measured by the visual analog scale, and incidence of side effects associated with the Difflam spray. This proposal will determine whether the use of Difflam spray is suitable to be implemented in local clinical setting and improve perioperative care.

DETAILED DESCRIPTION:
Postoperative sore throat (POST) after laryngeal mask airway (LMA) insertion is common, with reported incidences being as high as 40 - 60%. This is in spite of ongoing efforts to address this pertinent issue, including utilization of updated iterations of LMA devices, reduction of LMA cuff pressure, etc.. POST is an independent predictor of patient dissatisfaction following general anaesthesia and should be investigated further.

The cause of POST is multifactorial, with various mechanisms at play. A significant cause of POST is mechanical injury to the airway mucosa during airway instrumentation, leading to mucosal injury and inflammation. While the application of topical lidocaine on airway mucosa after surgery for analgesic relief may seem to be a possible solution, this may however, increase the risk of aspiration due to diminished cough reflex and swallowing ability. On the other hand, mouth gargles with analgesics may not provide immediate relief for POST as they require much cooperation from the patient that proves to be challenging in the immediate postoperative period.

The Difflam Forte Anti-Inflammatory Throat Spray is an over-the-counter medication indicated for temporary relief of painful mouth and throat conditions. It contains benzydamine hydrochloride (BH) 3 mg/mL, a non-steroidal anti-inflammatory agent (NSAID), and is recommended for adults to spray 2 to 4 times to the affected throat every 1.5 to 3 hours as needed. The effectiveness of benzydramine on alleviating sore throat has been well established in modern medicine. However, a spray formulation of this medication has not been utilized for this purpose yet. With the spray formulation, patient cooperation will not be required for effective delivery of BH medication - a critical factor in view of patient drowsiness post operation.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anaesthesiologists (ASA) physical status 1-2
2. Female patients having laryngeal mask airway (LMA) for airway management for surgery in KKH;
3. BMI < 40 kg/m2.

Exclusion Criteria:

1. Pregnant;
2. Pre-existing sore throat, or history of upper respiratory tract infection/ abnormalities, hypertension, chronic pain or anti-inflammatory drugs and antihypertensive treatment;
3. Allergies to benzydamine hydrochloride;
4. Symptomatic hiatus hernia;
5. Severe gastroesophageal reflux disease;
6. Contraindications to the use of LMA.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The participating site is a specialised hospital only for women and children.
Enrollment: 106 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative sore throat | 1 day; from the immediate and 4 hours postoperative recovery period
  Presence of postoperative sore throat (POST) during the immediate and 4 hours postoperative recovery period. At these two time points patients will be asked whether they have sore throat; and answering 'yes' will be considered as 'POST present'.

SECONDARY OUTCOMES:
Postoperative pain score | 1 day; from the immediate and 4 hours postoperative recovery period
  Pain score during the immediate and 4 hours postoperative recovery period after intervention (Visual analog scale 0-10) will be asked, with zero being no pain, and 10 being the worst pain possible.
Side effects | 1 day; from the immediate and 4 hours postoperative recovery period
  Presence of side effects during the immediate and 4 hours postoperative recovery period. At these two time points patients will be asked whether they have burning and/or stinging, dry mouth, cough, local numbness; and answering 'yes' will be considered as 'burning and/or stinging, dry mouth, cough, local numbness present'.

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
To be shared upon request